CLINICAL TRIAL: NCT00562250
Title: Pharmacokinetic Drug Interaction Study With Dapagliflozin and Glimepiride in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MB102-016
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Dapagliflozin
- Arm 2 (Active Comparator)
  Interventions: Drug: Glimepiride
- Arm 3 (Active Comparator)
  Interventions: Drug: Dapagliflozin + Glimepiride

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 20 mg, once daily, single dose
  Arms: Arm 1
Drug: Glimepiride — Tablets, Oral, 4 mg, once daily, single dose
  Arms: Arm 2
Drug: Dapagliflozin + Glimepiride — Tablets, Oral, Dapagliflozin 20 mg + Glimepiride 4 mg, once daily, single dose
  Arms: Arm 3

SUMMARY:
The purpose of the study is to determine the effect of glimepiride on dapagliflozin and the effect of dapagliflozin on glimepiride in healthy volunteers. In addition, the safety and tolerability of dapagliflozin with be assessed alone and while taking glimepiride

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with BMI of 18-32 kg/m2

Exclusion Criteria:

* Abnormal physical or lab findings
* Allergies to any sulfonylurea or related compounds

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration and exposure to glimepiride and dapagliflozin when administered alone and administered together | plasma concentrations will be measures as specified timepoints for 72 hours after each administred dose

SECONDARY OUTCOMES:
Measures of the plasma concentration of the active metabolite of glimepiride when administered alone or coadministered with glimepiride | for 72 hours after each administered dose
Recorded adverse events | for 72 hours after each administered dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Vicente López, Buenos Aires, Argentina

REFERENCES:
- See also: MB102-016 _CSR _synosis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3634&filename=MB102-016%20_CSR%20_synosis.pdf